CLINICAL TRIAL: NCT00050908
Title: Endothelial Function in HIV-Infected Subjects Prior To and After Starting a Potent Antiretroviral Regimen
Brief Title: Blood Vessel Function in HIV-Infected Patients Taking Anti-HIV Drugs
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: A5152s; ACTG A5152s; 10812 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2002-12-30; First posted 2003-01-01 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: Brachial Artery; Endothelium, Vascular; Vasodilation; Nitroglycerin; Reverse Transcriptase Inhibitors; HIV Protease Inhibitors; Drug Therapy, Combination; Ritonavir; efavirenz; lopinavir; stavudine; lamivudine; zidovudine; Treatment Naive
MeSH Terms: conditions — HIV Infections; Aneurysm

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a substudy of ACTG A5142. The purpose of this substudy is to evaluate blood vessel function in HIV-infected patients taking anti-HIV drugs.

DETAILED DESCRIPTION:
Endothelial dysfunction, assessed by measurement of brachial artery reactivity, is associated with coronary artery disease. Previous studies showed that patients taking HIV protease inhibitors (PIs) had a buildup of fatty deposits in their arteries and impaired flow-mediated vasodilation of the brachial artery, whereas endothelial function was normal in HIV-infected individuals not taking PIs. The effect of three different antiretroviral regimens on endothelial function in antiretroviral naïve HIV-infected patients will be examined in this substudy.

Patients in this substudy will have Brachial Artery Reactivity Tests (BARTs), which are painless ultrasound tests of an artery in the lower arm. Brachial artery reactivity will be measured at entry and at 4 and 24 weeks after patients are randomized to one of three open-label drug regimens in ACTG A5142. Brachial artery reactivity in response to two vasoactive stimuli (flow-mediated and nitroglycerin) will be assessed by measuring brachial artery diameter and flow velocity. Blood will be drawn at Weeks 4 and 24 for insulin and lipid tests. Patients will fast and refrain from tobacco and caffeine use for at least 8 hours prior to each study visit. For the duration of the substudy, patients will be asked not to change the amount of fruits, juices, antioxidants, and tea that they consume.

ELIGIBILITY:
Inclusion Criteria:

* Participation in ACTG A5142 .
* Able and willing to give written informed consent and to report current smoking status.
* Men who have been on stable testosterone replacement for at least 3 months prior to entry and plan to continue to receive a stable dose during the substudy may enroll. Men who have discontinued testosterone therapy must be off for at least 3 months to be eligible.
* Women receiving oral contraceptives, hormone replacement, or progestational derivatives must have been on stable regimens for at least 3 months prior to enrollment and must plan to remain on the same dose for the duration of the study. Women who have discontinued such therapy must be off for at least 3 months to be eligible.

Exclusion Criteria:

* Coronary heart disease, peripheral vascular disease, or cerebrovascular disease.
* Diabetes mellitus, with the exception of a previous history of gestational or steroid-induced diabetes mellitus within 12 weeks prior to substudy entry.
* Insulin-sensitizing agents such as metformin, pioglitazone, and rosiglitazone.
* Lipid-lowering drugs within 6 weeks prior to substudy entry.
* Systemic glucocorticoids, long-acting inhaled steroids, and certain anabolic steroids within 30 days prior to substudy entry.
* Uncontrolled hypertension.
* Heavy use of vitamin supplements.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca J. Torriani, M.D., Study Chair — University of California, San Diego
Locations (9):
- United States (9):
  - UCLA School of Med, Los Angeles, California
  - Univ of California, San Diego Antiviral Research Ctr, San Diego, California
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Chelsea Clinic, New York, New York
  - Univ of Cincinnati, Cincinnati, Ohio

REFERENCES:
- [Background] Stein JH, Klein MA, Bellehumeur JL, McBride PE, Wiebe DA, Otvos JD, Sosman JM. Use of human immunodeficiency virus-1 protease inhibitors is associated with atherogenic lipoprotein changes and endothelial dysfunction. Circulation. 2001 Jul 17;104(3):257-62. doi: 10.1161/01.cir.104.3.257. PMID 11457741
- [Background] Behrens G, Schmidt H, Meyer D, Stoll M, Schmidt RE. Vascular complications associated with use of HIV protease inhibitors. Lancet. 1998 Jun 27;351(9120):1958. doi: 10.1016/S0140-6736(98)26026-0. No abstract available. PMID 9654284
- [Background] Cleland SJ, Sattar N, Petrie JR, Forouhi NG, Elliott HL, Connell JM. Endothelial dysfunction as a possible link between C-reactive protein levels and cardiovascular disease. Clin Sci (Lond). 2000 May;98(5):531-5. PMID 10781383
- [Background] Henderson A. Endothelial dysfunction: a reversible clinical measure of atherogenic susceptibility and cardiovascular inefficiency. Int J Cardiol. 1997 Dec 1;62 Suppl 1:S43-8. doi: 10.1016/s0167-5273(97)00212-x. No abstract available. PMID 9464583
- [Background] Wolf K, Tsakiris DA, Weber R, Erb P, Battegay M; Swiss HIV Cohort Study. Antiretroviral therapy reduces markers of endothelial and coagulation activation in patients infected with human immunodeficiency virus type 1. J Infect Dis. 2002 Feb 15;185(4):456-62. doi: 10.1086/338572. Epub 2002 Jan 18. PMID 11865397
- [Result] Stein JH, Komarow L, Cotter BR, Currier JS, Dube MP, Fichtenbaum CJ, Gerschenson M, Mitchell CK, Murphy RL, Squires K, Parker RA, Torriani FJ; ACTG 5152s Study Team. Lipoprotein Changes in HIV-Infected Antiretroviral-Naive Individuals after Starting Antiretroviral Therapy: ACTG Study A5152s Stein: Lipoprotein Changes on Antiretroviral Therapy. J Clin Lipidol. 2008 Dec;2(6):464-471. doi: 10.1016/j.jacl.2008.08.442. PMID 19956354